CLINICAL TRIAL: NCT03733860
Title: Preservation of Penile Tumescence by Cavernous Tissue Preservation During Penile Prosthesis Implantation
Brief Title: Cavernous Tissue Preservation During Penile Prosthesis Implantation
Acronym: CTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham Zaazaa, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ2017
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; penile tumescence; cavernous tissue
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cavernous sparing group (Active Comparator)
  Interventions: Procedure: Cavernous tissue sparing penile prosthesis implantation; Procedure: Intracavernosal injection of alprostadil
- Conventional technique group (Other)
  Interventions: Procedure: Conventional penile prosthesis implantation

INTERVENTIONS:
Procedure: Cavernous tissue sparing penile prosthesis implantation — Beginning penile prosthesis implantation (Coloplast Titan USA) procedure after intracavenosal injection of PGE1 prostine.
  Arms: Cavernous sparing group
Procedure: Conventional penile prosthesis implantation — Beginning penile implant procedure (Coloplast Titan USA) without prior intracavernosal injection of PGE1 prostine
  Arms: Conventional technique group
Procedure: Intracavernosal injection of alprostadil — Intraoperative intracavernosal injection of alprostadil in the cavernous sparing group
  Arms: Cavernous sparing group

SUMMARY:
Spontaneous penile tumescence after penile prosthesis implantation has been previously reported as sporadically occurring during implant surgery. This study aims at systematically preserving residual erectile function, by the preservation of the patients' spontaneous penile tumescence by systematically sparing cavernous tissue during penile prosthesis implantation.

DETAILED DESCRIPTION:
Patients undergoing the cavernous tissue sparing penile implant procedure will be injected intraoperatively with 40µg alprostadil, a prostaglandin E1 agonist intracorporal injection (ICI). The procedure will begin as soon as maximal tumescence is attained.

In the cavernous sparing group, corporal dilation will be done solely with a size 8 dilator. The insertion of the dilator will be carefully inserted in what we call the path of least resistance. To determine the path of least resistance, the corporotomy is spread apart by pulling on previously set stay sutures. The path of least resistance is the plane with maximum outflow of blood from the intraoperatively pharmaceutically dilated and blood filled corpora cavernosa. This plane can also be anticipated with a preoperative penile duplex.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction not amenable to treatment by approved medical therapy

Exclusion Criteria:

* Erectile dysfunction amenable to treatment by approved medical therapy

Ages: 18 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cavernous tissue thickness postoperatively measured by ultrasound | 1 month

SECONDARY OUTCOMES:
Presence of spontaneous penile tumescence post operatively | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Adham Zaazaa, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaazaa A, Bayerle-Eder M, Elnabarawy R, Elbitar M, Mostafa T. Penile Hemodynamic Response to Phosphodiesterase Type V Inhibitors after Cavernosal Sparing Inflatable Penile Prosthesis Implantation: A Prospective Randomized Open-Blinded End-Point (PROBE) Study. Adv Urol. 2021 Jun 28;2021:5548494. doi: 10.1155/2021/5548494. eCollection 2021. PMID 34257646